CLINICAL TRIAL: NCT02359656
Title: Recent and Non United Odontoid Fractures: Clinical and Biomechanical Aspects
Brief Title: Recent and Non United Odontoid Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, Assoc. Prof. Priv. Doz. Dr. Patrick Platzer, PhD, MBA, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1127/2009
Record Dates: First submitted 2015-01-31; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Odontoid Process
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non operative treatment (Other): specif non operative treatment protocol
  Interventions: Other: non operative treatment for odontoid non unions
- operative treatment (Other): dorsal atlanto-axial C1-C2 Arthrodesis
  Interventions: Procedure: surgical treatment

INTERVENTIONS:
Procedure: surgical treatment — C1-C1 arthrodesis
  Arms: operative treatment
Other: non operative treatment for odontoid non unions — specific non operative treatment protocol
  Arms: non operative treatment

SUMMARY:
The purpose of this study was to determine the clinical and radiographic long - term results in geriatric patients who had undergone surgical or non - operative treatment of odontoid non - unions, with particular regards to late bony fusion, cervical spine motion, neurological sequela, and patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 65 years or older who had undergone surgical or non - operative management of odontoid non-unions were sorted and their dataset of follow - up monitoring was examined for completeness and accuracy. According to our inclusion criteria, patients with complete sets of collected data and a follow-up examination of at least five years after treatment of the non - union were finally enrolled in this study. Collected data included variables, such as age, gender, mechanism of injury, fracture type, associated injuries, presence and severity of primary neurological deficits, primary treatment, clinical and neurological outcome after primary treatment, methods of treatment, clinical and radiographic outcome after treatment of the non-union, as well as morbidity and mortality of the patients.

Exclusion Criteria:

Exclusion criteria for this study contain patients with previous or subsequent surgery at the cervical spine level, patients with incomplete data sets, as well as patients with penetrating mechanism of injury or congenital cervical spine anomalies. Incomplete data set was determined, if pertinent clinical or radiographic data of follow - up monitoring (e.g. documents of clinical findings or functional results, radiographs, CT-scanning, e.g.) were missing.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-01; Primary Completion 2013-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome (range of motion) and radiographic (bony fusion) long - term results in geriatric patients who had undergone surgical or non - operative treatment of odontoid non - unions. | follow up of at least 5 years

SECONDARY OUTCOMES:
Composite outcome measure consisting of multiple measures as late bony fusion, cervical spin, neurological sequalea | follow up of at least 5 years